CLINICAL TRIAL: NCT06261853
Title: Determining the Clinical IMPACT of 3D-CBCT Imaging in Comparison to 2D-OPG on Nerve Injuries During Wisdom Tooth Surgery
Brief Title: The Impact of 3D-CBCT Imaging on Nerve Injuries During Wisdom Tooth Surgery
Acronym: IMPACTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Zarqa University (Unknown); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2-081-23
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Inferior Alveolar Nerve Injuries; Impacted Third Molar Tooth
Keywords: nerve injury; wisdom tooth; impacted third molar; cone beam CT; OPG; CBCT; mandibular wisdom tooth
MeSH Terms: conditions — Mandibular Nerve Injuries | interventions — Radiography, Panoramic

STUDY DESIGN:
Intervention Model Description: Pragmatic, two-arm, single-blinded, randomised controlled trial designed to investigate the differences between 3D cone-beam computerised tomography (CBCT) and 2D orthopantomography (OPG) in reducing inferior alveolar nerve injuries during wisdom tooth surgery.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor) A single-blinded methodology will be employed due to the nature of the image-based investigation where the surgeon is required to utilise one imaging modality during the surgery. In order to eliminate any influence or bias on the outcomes and data obtained for the primary objective, both the subject (patient) and the study member who will do the follow-up call will be blinded to the imaging techniques used on the day of surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-CBCT Scan (Experimental): The surgeons will only utilise the 3D-CBCT scan of their patient during wisdom tooth surgery. The patient should observe no difference in their care in this arm of the trial on the day of surgery as they wouldn't typically be aware of which image was being viewed
  Interventions: Radiation: 3D-CBCT
- 2D-OPG X-ray (Active Comparator): The surgeons will only utilise the 2D-OPG X-ray of their patient during wisdom tooth surgery. The patient should observe no difference in their care in this arm of the trial on the day of surgery as they wouldn't typically be aware of which image was being viewed
  Interventions: Radiation: 2D-OPG

INTERVENTIONS:
Radiation: 3D-CBCT — CBCT provides a three-dimensional image of the hard tissue structures and their anatomical relationships such as the root of the wisdom tooth and the inferior dental canal. CBCT radiation doses are typically in the range of 60 microSv.
  Other Names: Cone Beam Computerised Tomography; Small Volume Cone Beam CT
  Arms: 3D-CBCT Scan
Radiation: 2D-OPG — An OPG provides a two-dimensional image of the hard tissue structures and their anatomical relationships such as the root of the wisdom tooth and the inferior dental canal. OPG radiation doses are typically in the range of 20 microSv.
  Other Names: Orthopantomography; Panoramic Dental X-ray
  Arms: 2D-OPG X-ray

SUMMARY:
The investigators aim to investigate if the additional information available from a 3D scan of the wisdom tooth can reduce the risk of nerve injury during wisdom tooth surgery compared to conventional 2D images.

Wisdom tooth surgery is a common surgical procedures that a significant proportion of the population will undergo. As with any other surgical procedure, there are potential complications, of which, injury to the nerve supplying feeling to the lip, chin, and tongue is the most significant. This can lead to persistent pain, tingling, or numbness that may impact a patient's ability to eat and function.

The risk of nerve injury during wisdom tooth surgery is assessed using X-ray images, which show the position of the nerve and tooth in the jawbone. 2D and 3D scans are used, which have their own advantages and disadvantages such as reduced cost and radiation dose with 2D or more information from 3D images, but it remains unclear which is better at reducing the risk of nerve injuries.

DETAILED DESCRIPTION:
This pragmatic clinical trial is a multi-centre, two-arm, single-blind randomised controlled trial.

The primary research question is:

1. Does the additional information provided by a 3D scan, over a 2D x-ray, reduce the number of nerve injuries occurring during wisdom tooth surgery.

The secondary objectives are:

1. Does the additional information provided by the 3D scan, over the 2D x-ray, reduce the operation time?
2. Does the additional information provided by the 3D scan, over the 2D x-ray, impact the number and type of complications occuring during wisdom tooth surgery?
3. Does the additional information provided by the 3D scan, over the 2D x-ray, impact the number and type of complications observed after wisdom tooth surgery?

The study intervention:

1. On the day of surgery, the surgeon will utilise only one imaging technique, either the 2D OPG or the 3D CBCT, during wisdom tooth surgery. The trial arm allocation will be noted on their operating list alongside the planned procedure details. Conventionally, surgeons would have access to both images and therefore, it is difficult to determine the relative impact of each on surgical outcomes. The patient should observe no difference in their care in either arm of the trial on the day of surgery as they wouldn't typically be aware of which image was being utilised.
2. Data will be collected peri-operatively by way of a proforma completed by the surgeon. If the surgeon feels the need to use the other imaging modality to which the patient is allocated, for example, to maintain standards of care, this will be recorded along with the reasons why. Operating time and intraoperative complications will also be documented for each surgical procedure.
3. One week after the surgery, participants will receive a follow-up phone call from a research team member, which should last no more than five minutes. They will be asked five 'yes/no' questions about their recovery. Typically, patients having wisdom tooth surgery are not routinely followed up after their surgery unless specifically requested by the surgeon, therefore, this could be seen as an improved level of care for most patients especially as the research team member will have access to the post-operative care instructions from the department and can ask a surgeon to contact the patient if requested or deemed necessary.
4. After the one-week postoperative telephone review, the participant will be discharged from the study even if they continue to receive post-operative care, as clinically indicated, from their surgeon. If the patient is subsequently listed for another wisdom tooth surgical procedure and still meets the inclusion criteria, they may be invited to enrol again in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals are seen in the Oral Surgery department with a 2D-OPG x-ray and a diagnosis of a mandibular wisdom tooth that requires surgical treatment.
2. Individuals requiring a 3D-CBCT to further assess the relationship between the wisdom tooth and the inferior alveolar nerve.
3. Individuals who are to undergo surgical treatment for their wisdom tooth regardless of the surgical approach (e.g. coronectomy or extraction) or the anaesthetic technique utilised.
4. Individuals without any pre-existing neurological deficit of cranial nerve V (trigeminal nerve) or medical conditions or medications that may cause changes in neurosensory function.
5. Individuals over the age of 16 and willing and able to provide valid informed consent for themselves.
6. Individuals with adequate English comprehension to read the written PIS and consent form and understand the follow-up call questions.
7. Individuals willing to provide contact details to allow a telephone follow-up call one week after their surgery.

Exclusion Criteria:

1. Individuals who do not have the capacity to consent for themselves.
2. Individuals taking medicines or having medical conditions and disorders that impair neurosensory function.
3. Individuals requiring wisdom tooth surgery to manage associated pathology such as cysts, fractures, or tumours where the pathological condition may interfere with the neurosensory function of the trigeminal nerve at 1 week post-operatively.
4. Individuals who are unable to read or speak English.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1292 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The number of patients reporting altered sensation in their lip and/or chin on the side of wisdom tooth surgery | one week after surgery
  The primary outcome measure is assessed by a series of yes/no questions asked during the follow-up call one week after the surgery.

SECONDARY OUTCOMES:
Surgical time | on the day of surgery
  Surgery duration from initiation of the procedure (knife to mucosa or start of elevation etc. not including anaesthesia time) to the completion of closure of the wound (not including post-op instructions etc.). This will be evaluated using data from the intraoperative surgeon's proforma which is completed by the surgeon on the day of surgery.
Planned surgical approach | on the day of surgery
  Surgical technique utilised either total removal (extraction) or intentional partial removal leaving the roots behind (coronectomy). This will be measured and reported using data from the intraoperative surgeon's proforma which is completed by the surgeon on the day of surgery.
Intraoperative complications | on the day of surgery
  The quantity and type of intraoperative complications (excessive bleeding, unintentional root retention, nerve exposure). This will be evaluated using data from the intraoperative surgeon's proforma which is completed by the surgeon on the day of surgery.
Postoperative Complications | one week after surgery
  The quantity and type of postoperative complications (altered sensation in the tongue, persistent swelling, and analgesia intake). This will be evaluated using data collected from a series of yes/no questions asked during the follow-up phone call.
Wisdom tooth impaction classification | on the day of surgery
  The classification of wisdom tooth impaction. This will be evaluated using data from the intraoperative surgeon's proforma which is completed by the surgeon on the day of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Lalli, BDS PhD, Study Chair — Institute of Dentistry, University of Aberdeen; Rahmeh Alhyari, BDS MFDS RCSEd, Study Director — Institute of Dentistry, University of Aberdeen
Locations (2):
- United Kingdom (2):
  - King'S College Hospital Nhs Foundation Trust, London, England
  - Aberdeen Dental Hospital, Aberdeen, Scotland

IPD SHARING:
Plan to Share IPD: No